CLINICAL TRIAL: NCT01351207
Title: The Effect of Eggs on Postprandial Metabolism: A Randomized, Controlled Crossover Pilot Study in Older, Overweight Adults
Brief Title: The Effect of Eggs on Postprandial Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB9795
Record Dates: First submitted 2011-04-27; First posted 2011-05-10 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
MeSH Terms: interventions — Eggs

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- pork sausages and hash brown potatoes plus eggs (Active Comparator)
  Interventions: Other: Eggs
- pork sausages and hash brown potatoes plus egg-free pudding (Placebo Comparator)
  Interventions: Other: Eggs
- pork sausages and hash brown potatoes (Placebo Comparator)
  Interventions: Other: Eggs

INTERVENTIONS:
Other: Eggs — Comparison of a high saturated fat/low fiber meal alone, with eggs, and with a protein/cholesterol matched egg-free pudding

SUMMARY:
The objective of this randomized, double-blinded, placebo-controlled, 3-way crossover pilot study is to determine whether eggs can favorably alter biomarkers of postprandial metabolism when included with other cooked breakfast foods typically selected by older Americans.

ELIGIBILITY:
Inclusion Criteria:

* Men & postmenopausal women, aged 50-70 years
* BMI 28-34 kg/m2

Exclusion Criteria:

* Cigarette smoking and/or nicotine replacement use
* Individuals taking estrogen
* Use of cholesterol-lowering medications
* Use of blood pressure-lowering medications
* Regular use of any stomach acid-lowering medications or laxatives (including fiber supplements)
* Cardiovascular (heart) disease
* Gastrointestinal disease
* Kidney disease
* Endocrine disease: including diabetes, untreated thyroid disease
* Rheumatoid arthritis
* Active treatment for any type of cancer, except basal cell carcinoma, within 1 year prior to study admission
* Systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 95 mmHg
* Regular use of oral steroids
* Regular daily intake of ≥ 2 alcoholic drinks
* Vegetarians
* Allergy to eggs
* Avoidance and/or intolerance of pork products
* No dietary supplements, including those containing any vitamins, minerals,herbs, plant concentrates (including garlic, gingko, St. John's wort) homeopathic remedies, probiotics, or fish oil (including cod liver oil), for one month prior to study admission

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Postprandial change in blood glucose concentration compared to placebo | 0-4 h
  Biomarkers of glucoregulation and insulin sensitivity, inflammation, lipid peroxidation, antioxidant activity, and satiety hormone production will be assessed in blood and urine

CONTACTS AND LOCATIONS:
Overall Officials: Diane L. McKay, PhD, Principal Investigator — Tufts Medical Center
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States